CLINICAL TRIAL: NCT07188779
Title: Impact of RADA16 Use on Outcomes Following Tonsillectomy in Children
Acronym: RADA16 for Ped
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Wayne Daniel Hsueh, MD, ASSOC PROF-CLIN, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2025001802
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain
Keywords: tonsillectomy; adenoidectomy; hemostasis; postop complications
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RADA16 (Active Comparator): Patients randomized to the treatment arm will undergo application of 2.5% RADA16 hydrogel to the tonsillar fossae following tonsillectomy using a sterile syringe tip applicator. The gel will be spread into a thin layer within the tonsillar fossae. The gel will be left to sit for 60 seconds. A suction device will then be used to remove any excess RADA16 hydrogel, leaving a thin layer of RADA16 over the tonsillar fossae.
  Interventions: Device: RADA16 hydrogel
- Control arm (No Intervention): Patients randomized to the control arm will not undergo application of RADA16 hydrogel following hemostasis with suction monopolar electrocautery.

INTERVENTIONS:
Device: RADA16 hydrogel — Application of 2.5% RADA16 hydrogel to the tonsillar fossae following tonsillectomy using a sterile syringe tip applicator. The gel will be spread into a thin layer within the tonsillar fossae. The gel will be left to sit for 60 seconds. A suction device will then be used to remove any excess RADA16 hydrogel, leaving a thin layer of RADA16 over the tonsillar fossae.
  Other Names: puragel
  Arms: RADA16

SUMMARY:
The purpose of the research is to determine if RADA16 (also known as PuraStat®, PuraGel®, or PuraSinus®) improves patient outcomes following pediatric tonsillectomy procedures. Researchers will compare application of device RADA16 to application of no device to see if RADA16 works to treat post tonsillectomy hemorrhage.Participants will:

Undergo tonsillectomy procedure. Receive and fill out a survey sent via email every 2 days following their procedure for 15 days, plus an additional survey on day 30, and track their symptoms.

DETAILED DESCRIPTION:
This is a prospective study evaluating the impact of intraoperative RADA16 application on the postoperative course following pediatric tonsillectomy as it relates to pain, bleeding, readmission, and use of a rescue analgesic (ex., oxycodone). We propose a randomized controlled trial whereby patients undergoing tonsillectomy would either receive a standard analgesic regimen (postoperative acetaminophen and NSAIDs plus oxycodone as a supplemental analgesic) versus intraoperative RADA16 application plus a standard analgesic regimen.

ELIGIBILITY:
Inclusion Criteria:

Children aged 3-17 years undergoing tonsillectomy +/- adenoidectomy CPT codes

* 42820 (Tonsillectomy and adenoidectomy; younger than age 12)
* 42821 (… age 12 or over)
* 42825 (Tonsillectomy; primary or secondary; younger than age 12)
* 42826 (… age 12 or over)
* 42830 (Adenoidectomy, primary; younger than age 12)
* 42831 (… age 12 or over)
* 42835 (Adenoidectomy; secondary; younger than age 12)
* 42836 (… age 12 or over)

Exclusion Criteria:

* Children with bleeding disorders or other hematologic malignancy or taking anticoagulant medications Developmental delay affecting pain reporting Children with known allergies to RADA16 components Children with prior tonsillectomy or tonsillotomy Children undergoing tonsillectomy with concern for cancer, Children taking opioids chronically prior to surgery, Anyone pregnant women, incarcerated individuals, children unable to speak English or Spanish

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | From enrollment to post-operative day 30.
  Pain assessed via the Wong Baker Faces scale. The primary outcome measure will be assessed via online survey on post-operative day one then subsequently every other day until post-operative day fifteen, with a final survey on day 30.

SECONDARY OUTCOMES:
Number of Participants with post-tonsillectomy hemorrhage who receive topical agents | From enrollment to post-operative day 30
  Number of Participants with post-tonsillectomy hemorrhage who receive topical agents for management of post tonsillectomy hemorrhage
Number of Participants with post-tonsillectomy hemorrhage who require a return to the operating room | From enrollment to post-operative day 30
  Number of Participants with post-tonsillectomy hemorrhage who require a return to the operating room for management of post tonsillectomy hemorrhage
Number of participants who require hospital readmission for post tonsillectomy hemorrhage management | From enrollment to post-operative day thirty
  Number of participants who require readmission for management of post tonsillectomy hemorrhage
Number of participants who require a rescue analgesic for management following tonsillectomy procedure | From enrollment to post-operative day 30
  Number of participants who use a rescue analgesic following their tonsillectomy procedure
Days participants take to resume their regular diet post operation | From enrollment to post-operative day 30
  Recording how many days it takes for participants to return to their regular diet post operation

IPD SHARING:
Plan to Share IPD: No
Determining if access to university data can be available for the study

REFERENCES:
- [Background] Mitchell RB, Archer SM, Ishman SL, Rosenfeld RM, Coles S, Finestone SA, Friedman NR, Giordano T, Hildrew DM, Kim TW, Lloyd RM, Parikh SR, Shulman ST, Walner DL, Walsh SA, Nnacheta LC. Clinical Practice Guideline: Tonsillectomy in Children (Update). Otolaryngol Head Neck Surg. 2019 Feb;160(1_suppl):S1-S42. doi: 10.1177/0194599818801757. PMID 30798778
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Pynnonen M, Brinkmeier JV, Thorne MC, Chong LY, Burton MJ. Coblation versus other surgical techniques for tonsillectomy. Cochrane Database Syst Rev. 2017 Aug 22;8(8):CD004619. doi: 10.1002/14651858.CD004619.pub3. PMID 28828761